

## **Informed Consent**

# INFORMED CONSENT/AUTHORIZATION FOR PARTICIPATION IN RESEARCH

Building a Diverse Biomedical Workforce Through Communication Across Difference 2019-1010

| Subtitle: Focus Groups | |
|-----------------------------|-----------------------------------|
| Study Chair: Carrie Cameron | |
| Participant's Name | Medical Record Number or Study ID |

This is an informed consent and authorization form for a research study. It includes a summary about the study. A more detailed description of procedures and risks is provided after the summary.

This research has been reviewed and approved by an Institutional Review Board (IRB - a committee that reviews research studies).

#### STUDY SUMMARY

You are being asked to take part in this part of the study because you recently participated in the "Communicating Across Difference" study workshops.

The goal of this research study is to investigate how STEM researchers communicate, including the role of mentors in building inclusive interpersonal communication skills. Researchers want to learn more about the factors that may help or block career goals and career persistence of researchers.

Study participation takes place with a study partner. Your study partner is your near-peer mentor if you are a research student. Your study partner is your research student mentee if you are a near-peer mentor. A "near-peer mentor" is defined as a PhD student, postdoctoral fellow, or instructor who has been assigned by a more senior faculty member or Principal Investigator as the day-to-day supervisor of a research student. If your study partner has not registered to participate, you may still participate by yourself.

# This is an investigational study.

You may benefit from this study by learning more about the effective communication skills in the STEM research environment. There may be no benefits for you in this study.

Your participation is completely voluntary. Before choosing to take part in this study, you should discuss with the study team any concerns you may have, including potential expenses and time commitment.

You can read a list of potential risks below in the Possible Risks section of this consent.

Your active participation in this phase of the study will be over after you complete the focus group.

There is no cost to you for taking part in this research study.

You may choose not to take part in this study.

## 1. STUDY DETAILS

In the current phase of this study, up to 40 research students and 40 near-peer mentors (PhD student, postdoctoral fellow, or instructor who has been assigned by a more senior faculty member or Principal Investigator as the day-to-day supervisor of a research student) will be enrolled in this study across the United States.

If you agree to take part in this study, you will participate in a 60-minute online focus group via videoconference. There will be up to 9 other participants in the group. The focus group discussion will be led by Christine Bell, Wisconsin Center for Education Research, University of Wisconsin-Madison, the CAD project's external collaborator. Topics discussed during the focus groups will be related to developing interpersonal communication skills in the research environment and their influence on mentoring relationships.

The focus group sessions will be audio recorded and transcribed (written down). Christine Bell will use the audio recording to ensure the accuracy of the transcript and then delete the audio. The audio recording will not be shared with any research team members. The transcript and any poll responses, chat, and whiteboard comments will also be saved.

#### **Focus Group Responses**

Your focus group responses will be used for research purposes only, and your responses will not be shared with any other study participant outside of your focus group. All responses collected during this study will be kept strictly confidential. Your responses will not be shared with anyone other than the research team. None of the researchers has a supervisory role over any of the participants. Your mentor or other

research team members will not have access to your answers. You are not required to disclose to your mentor whether you agreed to participate or not. You should not share your responses.

#### 2. POSSIBLE RISKS

You should discuss the risks of **focus group participation** with the study chair. The known risks are listed in this form, but they will vary from person to person. The focus group session may have questions, issues, and/or topics discussed that are sensitive in nature. Some questions may make you feel upset or uncomfortable. You may refuse to answer any question. If you have concerns during or after the focus groups, you are encouraged to contact the study chair.

Although every effort will be made to keep study data safe, there is a chance that your information could be lost or stolen. All study data will be stored in password-protected computers. There will be no personal identifying information connected to your answers. Once the study is over, the data without any identifying information will be published. At that time, the database with your contact information will no longer be active.

This study may involve unpredictable risks to the participants.

### 3. COSTS AND COMPENSATION

There are no plans to compensate you for any patents or discoveries that may result from your participation in this research.

As compensation for your time and effort, you will receive a \$20 Amazon gift card if you complete at least 90% of the focus group.

## **Additional Information**

- 4. You may ask the study chair (Dr. Carrie Cameron, at <a href="mailto:ccameron@mdanderson.org">ccameron@mdanderson.org</a> or 713-794-1476) any questions you have about this study. You may also contact the Chair of MD Anderson's Institutional Review Board (IRB a committee that reviews research studies) at 713-792-6477 with any questions that have to do with this study or your rights as a study participant.
- 5. You may choose not to take part in this study without any penalty or loss of benefits to which you are otherwise entitled. You may also withdraw from participation in this study at any time without any penalty or loss of benefits. If you withdraw from this study, you can still choose to be treated at MD Anderson.
- 6. This study or your participation in it may be changed or stopped without your consent at any time by the study chair, National Institute of General Medical Sciences, or the IRB of MD Anderson.

- 7. You will be informed of any new findings or information that might affect your willingness to continue taking part in the study and you may be asked to sign another informed consent and authorization form stating your continued willingness to participate in this study.
- 8. MD Anderson may benefit from your participation and/or what is learned in this study.
- 9. This study is sponsored and/or supported by: National Institute of General Medical Sciences.

# Future Research

## Data

Your personal information is being collected as part of this study. These data may be used by researchers at MD Anderson.

## Authorization for Use and Disclosure of Protected Health Information (PHI):

- A. During the course of this study, MD Anderson may be collecting and using your PHI. For legal, ethical, research, and safety-related reasons, the research team may share your PHI with:
  - The Office for Human Research Protections (OHRP)
  - The IRB and officials of MD Anderson
  - National Institute of General Medical Sciences, who is a sponsor or supporter of this study, and/or any future sponsors/supporters of the study
  - Study monitors and auditors who verify the accuracy of the information
  - Individuals who put all the study information together in report form

Study sponsors and/or supporters receive limited amounts of PHI. They may also view additional PHI in study records during the monitoring process. MD Anderson's contracts require sponsors/supporters to protect this information and limit how they may use it

The results of this research may be published in scientific journals or presented at medical meetings, but your identity will not be disclosed.

- B. Signing this consent and authorization form is optional but you cannot take part in this study if you do not agree and sign.
- C. MD Anderson will keep your PHI confidential when possible according to state and federal law. However, in some situations, health authorities could be required to reveal the names of participants.

Once disclosed outside of MD Anderson, federal privacy laws may no longer protect your PHI.

NCT05048290 Protocol 2019-1010 January 6, 2023 Page 5 of 6

D. The permission to use your PHI will continue indefinitely unless you withdraw your authorization in writing. Instructions on how to do this can be found in the MD Anderson Notice of Privacy Practices (NPP) or you may contact the Chief Privacy Officer of MD Anderson at 713-745-6636. If you withdraw your authorization, you will be removed from the study and the data collected about you up to that point can be used and included in data analysis. However, no further information about you will be collected.

NCT05048290 Protocol 2019-1010 January 6, 2023 Page 6 of 6

○ I DO wish to take part in this study.○ I DO NOT wish to take part in this study.